CLINICAL TRIAL: NCT04555356
Title: The Effect of Low Back Pain on Paraspinal Muscle Volumes in Adolescents
Brief Title: The Effect Of Low Back Pain on Paraspinal Muscles
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, fatma esra bahadir ulger, Principal investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRHRF
Record Dates: First submitted 2020-09-15; First posted 2020-09-18 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain
Keywords: adolescent; low back pain; lumbar disc herniation; paraspinal muscle; magnetic resonance imaging
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Low back pain is frequently seen in the adolescent age group, with a prevalence approaching that of the adult age group. The most common type is non-specific, self-limiting low back pain. LDH is rare in children and adolescents and generally presents with low back pain, with or without radiculopathy. The condition is usually unilateral (especially L4-5 or L5-S1). LDH is also mostly central type. Although there are many studies that have investigated the relationship between paraspinal muscle volumes and LBP and/or LDH in the adult age group, there are very few studies in adolescents. The principal aim of this study was to compare MF, ES, and PM volumes in adolescents with LBP with and without LDH using magnetic resonance imaging (MRI) and to determine whether these two conditions cause paraspinal muscle volume loss.

DETAILED DESCRIPTION:
The medical records of 229 patients who underwent MRI due to low back pain persisting for a minimum of twelve weeks between January 2018 and January 2020 were evaluated retrospectively. Twenty-four patients were excluded due to the presence of spondylolysis-listhesis, spinal alignment disorders including scoliosis and kyphosis, inflammatory diseases, or histories of spinal surgery and multilevel disc hernia. Two hundred five patients were finally enrolled. Age, gender, weight, and height were recorded, and BMI was calculated as weight/(height)². Participants were divided into two groups - with LDH (Group A) and without LDH (Group B). Right- and left-side PS, MF, and ES muscle volumes at intervertebral disc levels L4-L5 and L5-S1 were measured on Axial T2-weighted fast spin-echo sequences. All cross-sectional images at both levels (L4-5 and L5-S1) were generated by means of multiplanar reformat images. The muscles were identified by means of manual contouring at both disc levels. The fat components were then eliminated by application of the threshold technique, based on visual differences in pixel signal intensities. Volume measurement from cross-sectional images was based on the use of an automatic volume calculation tool.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-18
* LBP persisting for a minimum of twelve weeks

Exclusion Criteria:

* spondylolysis-listhesis
* spinal alignment disorders including scoliosis and kyphosis
* inflammatory diseases
* histories of spinal surgery
* multilevel disc hernia

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients (aged 10-17) with low back pain persisting for a minimum of twelve weeks
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of paraspinal muscle volumes in adolescents with LBP with and without LDH | 3 months
  Multifidus, erector spina and psoas major muscle volumes were measured using T2 weighted axial MR images at L4-5 and L5-S1 intervertebral disc levels.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Esra Bahadir Ulger, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Atasehir, Turkey (Türkiye)